## Prescription Opioid Management in Chronic Pain Patients: A Patient-Centered Activation Intervention

PI: Cynthia Campbell, PhD

PCORI Contract: IHS-1310-08734

Clinical Trials.gov Protocol ID: NCT02290223

Last updated: January 16, 2018

## **STATISTICAL PLAN**

Univariate analyses were used to obtain summary statistics for each outcome variable, and data transformation or categorization was completed as needed based on checks for normality. We compared baseline differences in outcome measures and patient characteristics between the two treatment arms. Using an intent-to-treat approach with the full sample, we also compared differences between intervention groups on outcome measures at 6 and 12 months, using chi-squared test for categorical measures (e.g., any use of portal tools) and t-test for continuous measures (e.g., PAM score). Tests for significance are not shown.